CLINICAL TRIAL: NCT06759922
Title: Clinical Efficacy and Safety of Glimepiride, Empagliflozin and Sitagliptin With Metformin in Type 2 Diabetes Mellitus: A Double and Triple Drug Therapy
Brief Title: Glimepiride, Empagliflozin, and Sitagliptin With Metformin for Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUHS-IRB # R-104/24
Record Dates: First submitted 2024-12-09; First posted 2025-01-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Metformin; Glimepiride; Sitagliptin; Empagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: Metformin + Glimepiride (Combination Therapy) (Active Comparator): Dual therapy (Fixed Dose Combination):
  Tab Metformin 500mg + Tab Glimepiride 2mg Dosage: One tablet per day for 90 days.
  Interventions: Drug: Tab Metformin + Tab Glimepiride
- Group B: Metformin + Empagliflozin (Combination Therapy) (Active Comparator): Dual therapy (Fixed Dose Combination):
  Tab Metformin 500mg + Tab Empagliflozin 12.5mg Dosage: One tablet per day for 90 days.
  Interventions: Drug: Tab Metformin + Tab Empagliflozin
- Group C: Metformin + Sitagliptin (Combination Therapy) (Active Comparator): Dual therapy (Fixed Dose Combination):
  Tab Metformin 500mg + Tab Sitagliptin 50mg Dosage: One tablet per day for 90 days.
  Interventions: Drug: Tab Metformin +Tab Sitagliptin
- Group D: Metformin + Empagliflozin + Sitagliptin (Combination Therapy) (Active Comparator): Triple Therapy:
  Tab Metformin 500mg + Tab Empagliflozin 12.5mg (Fixed Dose Combination) + Tab Sitagliptin 50mg Dosage: One tablet of each per day for 90 days.
  Interventions: Drug: Tab Metformin + Tab Empagliflozin + Tab Sitagliptin

INTERVENTIONS:
Drug: Tab Metformin + Tab Glimepiride — Tab Metformin 500mg+ Tab Glimepiride 2mg (FDC) once per orally for 90 days.
  Other Names: Tab Orinase-Met (2/500mg)
  Arms: Group A: Metformin + Glimepiride (Combination Therapy)
Drug: Tab Metformin + Tab Empagliflozin — Tab Metformin 500mg+Tab Empagliflozin 12.5mg (FDC) once per orally for 90 days.
  Other Names: Tab Jardy-Met (12.5/500mg)
  Arms: Group B: Metformin + Empagliflozin (Combination Therapy)
Drug: Tab Metformin +Tab Sitagliptin — Tab Metformin 500mg+Tab Sitagliptin 50mg (FDC) once per orally for 90 days.
  Other Names: Tab Sita-Met (50/500mg)
  Arms: Group C: Metformin + Sitagliptin (Combination Therapy)
Drug: Tab Metformin + Tab Empagliflozin + Tab Sitagliptin — Tab Metformin 500mg+Tab Empagliflozin 12.5mg (FDC) + Tab Sitagliptin 50mg once per orally for 90 days.
  Other Names: Tab Jardy-Met (12.5/500mg) + Tab Sita 50mg
  Arms: Group D: Metformin + Empagliflozin + Sitagliptin (Combination Therapy)

SUMMARY:
This clinical trial aims to evaluate and compare the clinical efficacy and safety of Glimepiride, Empagliflozin, and Sitagliptin with Metformin in newly diagnosed Type 2 Diabetes Mellitus patients.

The study will involve 172 participants, aged 30-55, enrolled at the National Medical Centre, Karachi, Pakistan. The study involves four groups, subjects will receive following treatment: Group A will receive Tab Metforrmin 500mg + Tab Glimepiride 2mg (FDC) , Group B Tab Metforrmin 500mg + Tab Empagliflozin 12.5mg (FDC), Group C Tab Metforrmin 500mg + Tab Sitagliptin 50mg (FDC) and Group D Tab Metformin 500mg + Tab Empagliflozin 12.5mg (FDC) + Tab Sitagliptin 50mg per orally, once daily for 90 days. Safety and efficacy will be assessed through anthropometric measurements and lab investigations at baseline, 6 weeks, and 12 weeks, with weekly monitoring of blood sugar levels. The total duration of the study will be 6 months, with a 3-month individual treatment period.

DETAILED DESCRIPTION:
To evaluate and compare the clinical efficacy and safety of Glimepiride, Empagliflozin and Sitagliptin with Metformin in Type 2 Diabetes Mellitus: A double and triple drug therapy.

Newly diagnosed males and females with type 2 diabetes mellitus having age between 30 to 55 yrs presenting in diabetic OPD of National Medical Centre Karachi Pakistan.

This clinical trial will be conducted on 135±37=172 newly diagnosed cases of Type 2 Diabetes Mellitus in the National Medical Centre after approval from IRB of Bahria University Health Sciences Campus Karachi. Patients will be enrolled after taking written informed consent. The study design is Randomized open label, parallel arms, clinical trial. They will be randomized into four groups using a sealed envelop method and a non-probability consecutive sampling technique. Total sample size is 135 with 33 patients in each group. However, investigator will work on 172 subjects 43 in each group. Group A will receive fixed drug combination (FDC) of Tab Metforrmin 500mg + Tab Glimepiride 2mg, Group B Tab Metforrmin 500mg + Tab Empagliflozin 12.5mg, Group C Tab Metforrmin 500mg + Tab Sitagliptin 50mg and Group D Tab Metformin 500mg + Tab Empagliflozin 12.5mg (FDC) + Tab Sitagliptin 50mg per orally, once daily for 90 days.

Complete safety profile parameters and analysis, will be done at baseline, week 6 and week 12 in addition to the following:

Baseline= Anthropometric measurements (weight, height, BMI, waist, hip circumference, waist to hip ratio, neck circumference) and all Lab investigation (Glycemic profile including Fasting Blood Sugar, Random Blood Sugar, HbA1c), (Lipid profile TC mg/dL, TG mg/dL, HDL mg/dL, LDL mg/dL, VLDL mg/dL), safety profile (blood (CBC) renal (Serum urea, Serum creatinine, Glomerular Filtration Rate, Urine for Microalbumin) hepatic (Alanine Transaminase, AspartateAminotransferase) and cardiac (Triglycerides, High Density Lipoprotein, Uric Acid).

FBS & RBS on weekly basis Day 45= Anthropometric measurements (weight, height, BMI, waist, hip circumference, waist to hip ratio, neck circumference) and lab investigations (only FBS or RBS) will be done. Adverse events (nausea, vomiting, diarrhea, hypoglycemia, weight gain, constipation, headache, urinary tract infection, flu like symptoms and any others) Day 90= Anthropometric measurements (weight, height, BMI, waist, hip circumference, waist to hip ratio, neck circumference), all Lab investigation (Glycemic profile including Fasting Blood Sugar, Random Blood Sugar, HbA1c), (Lipid profile TC mg/dL, TG mg/dL, HDL mg/dL, LDL mg/dL, VLDL mg/dL), safety profile (blood (CBC) renal (Serum urea, Serum creatinine, Glomerular Filtration Rate, Urine for Microalbumin) hepatic (Alanine Transaminase, AspartateAminotransferase) and cardiac (Triglycerides, High Density Lipoprotein, Uric Acid). Adverse events ( nausea, vomiting, hypoglycemia, weight gain, diarrhea, constipation, headache, urinary tract infection, flu like symptoms and any others)

Individual study period will be 3 months. Total duration of study will be 6 months.

Expected outcome of the study will be:

1. Clinical Efficacy Evaluation:

   Improvement is expected regarding anthropometric measures such as weight, BMI, hip circumference, and waist circumference, they will be measured to track changes in body composition.

   Assessment of glycemic indicators, including glycated hemoglobin (HbA1c), random blood sugar (RBS), and fasting blood sugar (FBS), in order to gauge progress in glucose regulation.

   To detect any positive changes in lipid levels, lipid profile parameters such as total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides will be done and analyzed.
2. Comparison of Clinical Efficacy:

   Evaluation of the effects on anthropometric, glycemic, and lipid profile parameters of the effectiveness of four combination treatments (Metformin + Glimepiride, Metformin +Empagliflozin, Metformin + Sitagliptin, and Metformin + Sitagliptin + Empagliflozin). Determination of which drug combination regimen will be better based on the results observed.
3. Assesment of Adverse Effects:

   Monitoring and recording of side effects, such as genitourinary infections, gastrointestinal symptoms, and other reported side effects, related to each drug combination regimen. A comparison of the various treatment groups' adverse effect rates and severity.
4. Safety Evaluation:

To ensure the safety of the combination drug regimens, safety profiles will be evaluated using blood parameters, renal function tests, hepatic function tests, and cardiac parameters.

For point #2,3 &4, to come up with a best drug combination regimen for our type2 diabetics.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 30-55yrs
* HbA1c = ≥ 8.5 <10 mmol/mol (ADA. 2018)
* BMI >18.5- <29.9 (WHO Asian Criteria)
* Treatment naïve patients
* With / without dyslipidemia.

Exclusion Criteria:

* HbA1c >10 mmol/mol
* BMI > 30
* Pregnancy or lactation
* Systemic diseases such as: hypertension, thyroid, liver, renal diseases etc.
* Known allergy or intolerance to Metformin, Glimepiride, Sitagliptin or Empagliflozin.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | 3 months
  Change in HbA1c levels in %

SECONDARY OUTCOMES:
Secondary Outcome | 3months
  1. Change in BMI (weight and height will be combined to report BMI in kg/m^2)
  2. Change in Lipid Profile in mg/dL
  3. Incidence of Treatment-Emergent Adverse Events Metformin (Diarrhea) Glimepiride (Weight gain, Hypoglycemia) Empagliflozin (Urinary incontinence, Genitourinary infections) Sitagliptin (Gastrointestinal symptoms, Pancreatitis, Upper respiratory tract infections)

CONTACTS AND LOCATIONS:
Overall Officials: Saima Chandio, MBBS, Principal Investigator — Bahria University Islamabad
Locations (1):
- National Medical Center, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
All Data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD data will become accessible one year after publication and will remain available indefinitely.
Access Criteria: All the data will be accessible to everyone.

REFERENCES:
- [Background] Ahmed M, Saeed A, Khan MZ, Javaid SZ, Aslam F, Dar SI. A Comparison of the Effects of Empagliflozin and Sitagliptin, When Combined With Metformin, on Lipid Levels in Patients with Type 2 Diabetes: A Clinical Investigation. Cureus. 2023 Sep 5;15(9):e44709. doi: 10.7759/cureus.44709. eCollection 2023 Sep. PMID 37809225
- [Background] Davies MJ, Aroda VR, Collins BS, Gabbay RA, Green J, Maruthur NM, Rosas SE, Del Prato S, Mathieu C, Mingrone G, Rossing P, Tankova T, Tsapas A, Buse JB. Management of hyperglycaemia in type 2 diabetes, 2022. A consensus report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetologia. 2022 Dec;65(12):1925-1966. doi: 10.1007/s00125-022-05787-2. Epub 2022 Sep 24. PMID 36151309
- [Background] Dominguez Rieg JA, Rieg T. What does sodium-glucose co-transporter 1 inhibition add: Prospects for dual inhibition. Diabetes Obes Metab. 2019 Apr;21 Suppl 2(Suppl 2):43-52. doi: 10.1111/dom.13630. PMID 31081587
- [Background] ElSayed NA, Aleppo G, Aroda VR, Bannuru RR, Brown FM, Bruemmer D, Collins BS, Hilliard ME, Isaacs D, Johnson EL, Kahan S, Khunti K, Leon J, Lyons SK, Perry ML, Prahalad P, Pratley RE, Seley JJ, Stanton RC, Gabbay RA, on behalf of the American Diabetes Association. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Care in Diabetes-2023. Diabetes Care. 2023 Jan 1;46(Suppl 1):S140-S157. doi: 10.2337/dc23-S009. PMID 36507650
- [Background] Huang J, Liu X, Wei Y, Li X, Gao S, Dong L, Rao X, Zhong J. Emerging Role of Dipeptidyl Peptidase-4 in Autoimmune Disease. Front Immunol. 2022 Mar 4;13:830863. doi: 10.3389/fimmu.2022.830863. eCollection 2022. PMID 35309368
- [Background] Hur KY, Moon MK, Park JS, Kim SK, Lee SH, Yun JS, Baek JH, Noh J, Lee BW, Oh TJ, Chon S, Yang YS, Son JW, Choi JH, Song KH, Kim NH, Kim SY, Kim JW, Rhee SY, Lee YB, Jin SM, Kim JH, Kim CH, Kim DJ, Chun S, Rhee EJ, Kim HM, Kim HJ, Jee D, Kim JH, Choi WS, Lee EY, Yoon KH, Ko SH; Committee of Clinical Practice Guidelines, Korean Diabetes Association. 2021 Clinical Practice Guidelines for Diabetes Mellitus of the Korean Diabetes Association. Diabetes Metab J. 2021 Jul;45(4):461-481. doi: 10.4093/dmj.2021.0156. Epub 2021 Jul 30. PMID 34352984
- [Background] Janani L, Bamehr H, Tanha K, Mirzabeigi P, Montazeri H, Tarighi P. Effects of Sitagliptin as Monotherapy and Add-On to Metformin on Weight Loss among Overweight and Obese Patients with Type 2 Diabetes: A Systematic Review and Meta-Analysis. Drug Res (Stuttg). 2021 Nov;71(9):477-488. doi: 10.1055/a-1555-2797. Epub 2021 Aug 13. PMID 34388848
- [Background] Kim HJ, Noh JH, Moon MK, Choi SH, Ko SH, Rhee EJ, Hur KY, Jeong IK. A Multicenter, Randomized, Open-Label Study to Compare the Effects of Gemigliptin Add-on or Escalation of Metformin Dose on Glycemic Control and Safety in Patients with Inadequately Controlled Type 2 Diabetes Mellitus Treated with Metformin and SGLT-2 Inhibitors (SO GOOD Study). J Diabetes Res. 2024 Jan 5;2024:8915591. doi: 10.1155/2024/8915591. eCollection 2024. PMID 38223523
- [Background] Lovic D, Piperidou A, Zografou I, Grassos H, Pittaras A, Manolis A. The Growing Epidemic of Diabetes Mellitus. Curr Vasc Pharmacol. 2020;18(2):104-109. doi: 10.2174/1570161117666190405165911. PMID 30961501
- [Background] Magkos F, Hjorth MF, Astrup A. Diet and exercise in the prevention and treatment of type 2 diabetes mellitus. Nat Rev Endocrinol. 2020 Oct;16(10):545-555. doi: 10.1038/s41574-020-0381-5. Epub 2020 Jul 20. PMID 32690918
- [Background] Packer M, Anker SD, Butler J, Filippatos G, Ferreira JP, Pocock SJ, Sattar N, Brueckmann M, Jamal W, Cotton D, Iwata T, Zannad F; EMPEROR-Reduced Trial Committees and Investigators. Empagliflozin in Patients With Heart Failure, Reduced Ejection Fraction, and Volume Overload: EMPEROR-Reduced Trial. J Am Coll Cardiol. 2021 Mar 23;77(11):1381-1392. doi: 10.1016/j.jacc.2021.01.033. PMID 33736819
- [Background] Shin H, Schneeweiss S, Glynn RJ, Patorno E. Trends in First-Line Glucose-Lowering Drug Use in Adults With Type 2 Diabetes in Light of Emerging Evidence for SGLT-2i and GLP-1RA. Diabetes Care. 2021 Aug;44(8):1774-1782. doi: 10.2337/dc20-2926. Epub 2021 Jun 18. PMID 34385345
- [Background] Tomic D, Shaw JE, Magliano DJ. The burden and risks of emerging complications of diabetes mellitus. Nat Rev Endocrinol. 2022 Sep;18(9):525-539. doi: 10.1038/s41574-022-00690-7. Epub 2022 Jun 6. PMID 35668219
- [Background] Uusitupa M, Schwab U. Evolving Nutritional Therapy for Diabetes Mellitus. Nutrients. 2020 Feb 6;12(2):423. doi: 10.3390/nu12020423. PMID 32041141